CLINICAL TRIAL: NCT03362476
Title: Computer-based Alcohol Reduction Intervention for Alcohol-using HIV/HCV+ Russian Women in Clinical Care
Brief Title: Computer-based Intervention for Alcohol-using HIV/HCV+ Women
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: New York University (Other)
Collaborators: National Institute on Alcohol Abuse and Alcoholism (NIAAA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: IRB00094637; R01AA025882-01 (NIH)
Record Dates: First submitted 2017-11-30; First posted 2017-12-05 (Actual); Results first posted 2025-01-09 (Actual); Last update posted 2025-01-09 (Actual); Status verified 2022-09

CONDITIONS: Human Immunodeficiency Virus; Hepatitis C; Alcohol Abuse
Keywords: Human Immunodeficiency Virus; Hepatitis C; Computer Intervention; Alcoholism; Women; Russia
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome; Hepatitis C; Alcoholism | interventions — Ethanol; Standard of Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Computer-based alcohol reduction intervention + Clinician-delivered brief MET counseling (Experimental): Brief, computer-based, alcohol reduction intervention based on motivational enhancement therapy (MET) tailored for HIV/HCV co-infected women who used alcohol.
  Clinician-based MET counseling plus standard-of-care (SOC) for current substance users.
  Interventions: Behavioral: Computer-based alcohol reduction intervention; Behavioral: Brief clinician-delivered MET; Behavioral: Standard of care
- Clinician-delivered brief MET counseling (Active Comparator): Clinician-based brief MET counseling plus standard-of-care (SOC) for current substance users. only
  Interventions: Behavioral: Brief clinician-delivered MET; Behavioral: Standard of care

INTERVENTIONS:
Behavioral: Computer-based alcohol reduction intervention — Brief computer-based version of motivation enhancement therapy (MET) used in conjunction with clinician-delivered MET and standard clinical care for current substance users. Modules and follow up assignments focus on key concepts in substance use, including cravings, problem solving and decision making skills. The multimedia presentation, based on elementary level computer learning games, requires no previous experience with computers.The intervention was adapted to be linguistically, gender- and HIV/HCV-appropriate for Russian women living with HIV/HCV.
  Arms: Computer-based alcohol reduction intervention + Clinician-delivered brief MET counseling
Behavioral: Brief clinician-delivered MET — Clinician-delivered MET used in conjunction with standard clinical care for current substance users. The brief intervention is focused on goals, cravings, problem-solving and decision-making. The intervention was adapted to be linguistically, gender- and HIV/HCV-appropriate for Russian women living with HIV/HCV.
Behavioral: Standard of care — Clinicians ask about substance use and provide evidence-based recommendations promoting abstinence.

SUMMARY:
The study harnessed the multidisciplinary expertise of our research team to develop a brief, computer-based, alcohol reduction intervention tailored for HIV/HCV co-infected women and evaluate its efficacy. The intervention, if effective, may be an efficient and cost-effective alcohol reduction strategy, that is scalable and can be readily disseminated and integrated in clinical care at other AIDS Centres in Russia to enhance women's health and reduce HIV/HCV transmission risk.

DETAILED DESCRIPTION:
Women co-infected with human immunodeficiency viruses (HIV) and Hepatitis C (HCV) are at elevated risk for adverse health outcomes associated with alcohol use. Evidence-based alcohol reduction interventions for this vulnerable population are limited. To address this gap, the study harnessed the multidisciplinary expertise and experience of collaborative Russian-U.S. research team to develop a brief, computer-based, alcohol reduction intervention tailored for HIV/HCV co-infected women and evaluate its efficacy. The study was conducted in three sequential stages: (1) Adaptation, (2) Implementation, and (3) Evaluation. Participants will be randomized to one of two conditions: (1) adapted computer-based alcohol reduction intervention PLUS PLUS provider-delivered brief motivational counseling, or (2) provider-delivered brief motivational counseling. The trial design and analysis provide an appropriate conceptual and methodological framework to assess the efficacy of the computer-based intervention. The intervention, if effective, may be an efficient and cost-effective alcohol reduction strategy that is scalable and can be readily disseminated and integrated in clinical care at other AIDS Centres in Russia to enhance women's health and reduce HIV/HCV transmission risk.

ELIGIBILITY:
Inclusion Criteria:

* female;
* receiving HIV medical care at the AIDS Center;
* chart-documented HIV and chronic HCV infection;
* currently prescribed an antiretroviral (ARV) regimen;
* medically, cognitively, and psychologically capable of study participation;
* laboratory-confirmed recent alcohol use as detected by a Ethylglucuronide (EtG) analysis or self-reported alcohol use

Exclusion Criteria:

* not identifying as biological female
* not HIV and HCV positive
* no laboratory-confirmed or self-reported
* not willing to participate in the trial
* not able to participate in the trial due to medical, cognitive, or psychological issues

Ages: 21 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes
Enrollment: 200 (Actual)
Dates: Start 2018-01-03 (Actual); Primary Completion 2022-02-28 (Actual); Study Completion 2022-02-28 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ralph J Diclemente, PhD, Principal Investigator — New York University
Locations (2):
- New York University, New York, New York, United States
- North West District AIDS Center, Saint Petersburg, Russia

IPD SHARING:
Plan to Share IPD: Yes
Deidentified (IPD) collected in this study will be made available to other researchers.
Supporting Information: Study Protocol, SAP
Time Frame: Will be shared upon request by investigators
Access Criteria: Request from researcher to the PIs for use explaining nature of use; use must be for research purposes; willingness to share eventual abstracts and/or publications with the PIs

REFERENCES:
- [Background] DiClemente RJ, Brown JL, Capasso A, Revzina N, Sales JM, Boeva E, Gutova LV, Khalezova NB, Belyakov N, Rassokhin V. Computer-based alcohol reduction intervention for alcohol-using HIV/HCV co-infected Russian women in clinical care: study protocol for a randomized controlled trial. Trials. 2021 Feb 17;22(1):147. doi: 10.1186/s13063-021-05079-x. PMID 33596972
- [Background] Khalezova NB, Capasso A, Boeva EV, Gutova LV, Rassokhin VV, Neznanov NG, Belyakov NA, Brown JL, DiClemente RJ. Situational and motivational factors associated with unhealthy alcohol use among Russian women with HIV and hepatitis C Virus co-infection. Drug Alcohol Depend Rep. 2022 Jun;3:100053. doi: 10.1016/j.dadr.2022.100053. Epub 2022 Apr 14. PMID 35783993
- [Background] Brown JL, Anastasakis I, Revzina N, Capasso A, Boeva E, Rassokhin V, Crusey A, Sales JM, Hitch A, Renfro T, DiClemente RJ. Development and Cultural Adaptation of a Computer-Delivered and Multi-Component Alcohol Reduction Intervention for Russian Women Living with HIV and HCV. J Int Assoc Provid AIDS Care. 2021 Jan-Dec;20:23259582211044920. doi: 10.1177/23259582211044920. PMID 34668412

RESULTS

PARTICIPANT FLOW:
Groups:
- Computer-based Alcohol Reduction Intervention + Clinician-delivered Brief MET Counseling: Brief, computer-based, alcohol reduction intervention based on motivational enhancement therapy (MET) tailored for HIV/HCV co-infected women who used alcohol.
  Clinician-based MET counseling plus standard-of-care (SOC) for current substance users.
  Computer-based alcohol reduction intervention: Brief computer-based version of motivation enhancement therapy (MET) used in conjunction with clinician-delivered MET and standard clinical care for current substance users. Modules and follow up assignments focus on key concepts in substance use, including cravings, problem solving and decision making skills. The multimedia presentation, based on elementary level computer learning games, requires no previous experience with computers.The intervention was adapted to be linguistically, gender- and HIV/HCV-appropriate for Russian women living with HIV/HCV.
  Brief clinician-delivered MET: Clinician-delivered MET used in conjunction with standard clinical care for current substance users. The brief intervention is focused on goals, cravings, problem-solving and decision-making. The intervention was adapted to be linguistically, gender- and HIV/HCV-appropriate for Russian women living with HIV/HCV.
  Standard of care: Clinicians ask about substance use and provide evidence-based recommendations promoting abstinence.
- Clinican-delivered Brief MET Counseling: Clinician-based brief MET counseling plus standard-of-care (SOC) for current substance users. only
  Brief clinician-delivered MET: Clinician-delivered MET used in conjunction with standard clinical care for current substance users. The brief intervention is focused on goals, cravings, problem-solving and decision-making. The intervention was adapted to be linguistically, gender- and HIV/HCV-appropriate for Russian women living with HIV/HCV.
  Standard of care: Clinicians ask about substance use and provide evidence-based recommendations promoting abstinence.
Period: Overall Study
Arm/Group | Computer-based Alcohol Reduction Intervention + Clinician-delivered Brief MET Counseling | Clinican-delivered Brief MET Counseling
Started | 98 | 102
Completed | 98 | 101
Not Completed | 0 | 1
Not completed — Withdrawal by Subject | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Computer-based Alcohol Reduction Intervention + Clinician-delivered Brief MET Counseling | Clinican-delivered Brief MET Counseling | Total
Number analyzed (Participants) | 98 | 102 | 200
Age, Continuous [Mean (Standard Deviation); unit: years] | 35 (3.7) | 35 (4.0) | 35 (3.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 98 | 102 | 200
  Male | 0 | 0 | 0
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  Russia | 98 | 102 | 200
Percentage of Women Who Test Ethyl Glucuronide (EtG) Negative [Count of Participants; unit: Participants] — Percentage of women who test ethyl glucuronide (EtG) negative at baseline before randomization. Ethyl glucuronide will be measured in urine, with a sample taken at point-of-care at baseline. The definition of EtG negative is <500ng/mL. A dichotomous score will be created with participants testing EtG negative at baseline assigned a 0 and participants testing EtG positive at baseline assigned a 1.
  Participants | 34 | 33 | 67

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Women Who Test Ethyl Glucuronide (EtG) Negative
Description: Percentage of women who test ethyl glucuronide (EtG) negative will be estimated to evaluate the efficacy of the adapted computer-based alcohol reduction intervention condition, relative to standard of care condition. Ethyl glucuronide will be measured in urine, with a sample taken at point-of-care at baseline and follow-ups. The definition of EtG negative is <500ng/mL. A dichotomous score will be created for times 3, 6, and 9-months post baseline, with participants testing EtG negative over the three time points assigned a 0 and participants testing EtG positive at any of the three follow-up points assigned a 1.
Time Frame: 3-, 6-, and 9-month post-baseline
Measure: Count of Participants; unit: Participants
Arm/Group | Computer-based Alcohol Reduction Intervention + Clinician-delivered Brief MET Counseling | Clinican-delivered Brief MET Counseling
Number analyzed (Participants) | 98 | 102
Participants | 93 | 99

2. Secondary Outcome: Percentage of Women Who Test Phosphatidylethanol (PEth) Negative (<= 8 ng/mL)
Description: Percentage of women who test PEth negative (<= 8 ng/mL) will be estimated to evaluate the efficacy of the adapted computer-based alcohol reduction intervention condition, relative to standard of care condition.
Time Frame: 9-month post-baseline
Population: Number of participants who had PEth<8ng/mL at 9-months post-baseline
Measure: Number; unit: participants
Arm/Group | Computer-based Alcohol Reduction Intervention + Clinician-delivered Brief MET Counseling | Clinician-delivered Brief MET Counseling
Number analyzed (Participants) | 98 | 101
participants | 44 | 43

3. Secondary Outcome: Percentage of Participants in the Intervention Group With an Undetectable HIV Viral Load Compared to the Percentage of Women in the Control Group With an Undetectable Viral Load
Description: HIV viral load (VL) will be measured by testing blood to evaluate HIV disease progression. The measure is the number of participants with an undetectable viral load (<200 HIV copies per milliliter of blood.). A dichotomous measure is created by which any participant who has an undetectable viral load at 9-month post-baseline is assigned a 0 and any participant with a detectable viral load at that time point is assigned a 1.
Time Frame: 9-month post-baseline
Measure: Count of Participants; unit: Participants
Arm/Group | Computer-based Alcohol Reduction Intervention + Clinician-delivered Brief MET Counseling | Clinican-delivered Brief MET Counseling
Number analyzed (Participants) | 98 | 101
Participants | 16 | 26

4. Secondary Outcome: CD4 Cell Count
Description: CD4 count will be measured at 9-months post-baseline and compared between intervention groups. CD4 is measured as the number of CD4 cells per cubic mm of blood.
Time Frame: 9-month post-baseline
Measure: Mean (Standard Deviation); unit: CD4 cells/mm
Arm/Group | Computer-based Alcohol Reduction Intervention + Clinician-delivered Brief MET Counseling | Clinician-delivered Brief MET Counseling
Number analyzed (Participants) | 98 | 101
CD4 cells/mm | 532.1 (155.1) | 502.9 (111.4)

5. Secondary Outcome: Count of Women With a Severe FibroTest Score (3-4) at 9-month Post Baseline
Description: FibroTest, is a biomarker test that uses the results of six blood serum tests to generate a score that is correlated with the degree of liver damage. It combines α2-macroglobulin, haptoglobin, γ-glutamyl transpeptidase, apolipoprotein A1, alanine transaminase, and total bilirubin. FibroTest is scored on a scale of 0-4 depending on severity: 0-1 being mild liver damage; 1-2 being moderate; and 3-4 being severe damage. This outcome presents the count of women with a severe FibroTest score (3-4) at 9-months post baseline.
Time Frame: 9-month post-baseline
Measure: Count of Participants; unit: Participants
Arm/Group | Computer-based Alcohol Reduction Intervention + Clinician-delivered Brief MET Counseling | Clinician-delivered Brief MET Counseling
Number analyzed (Participants) | 98 | 101
Participants | 24 | 22

6. Secondary Outcome: Liver Stiffness
Description: FibroScan - imaging modality - will be used to measure liver stiffness at 9-months post-baseline and compared by intervention group. Liver stiffness is diagnosed by a medical specialist.
Time Frame: 9-month post-baseline
Population: Liver stiffness at to 9-month post-baseline (Yes)
Measure: Count of Participants; unit: Participants
Arm/Group | Computer-based Alcohol Reduction Intervention + Clinician-delivered Brief MET Counseling | Clinician-delivered Brief MET Counseling
Number analyzed (Participants) | 98 | 101
Participants | 84 | 90

ADVERSE EVENTS:
Time Frame: 9 months
Arm/Group | Computer-based Alcohol Reduction Intervention + Clinician-delivered Brief MET Counseling | Clinican-delivered Brief MET Counseling
All-Cause Mortality (participants affected / at risk) | 0/98 | 0/102
Serious Adverse Events (participants affected / at risk) | 0/98 | 0/102
Other Adverse Events (participants affected / at risk) | 0/98 | 0/102

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2021-02-01): https://cdn.clinicaltrials.gov/large-docs/76/NCT03362476/Prot_SAP_000.pdf
  • Informed Consent Form (2019-09-05): https://cdn.clinicaltrials.gov/large-docs/76/NCT03362476/ICF_001.pdf